CLINICAL TRIAL: NCT05873543
Title: The Effect of a Smartphone-assisted Hybrid Cardiac Rehabilitation Program in Patients With Heart Failure.
Acronym: SHCR-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202302009RINC
Record Dates: First submitted 2023-05-01; First posted 2023-05-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: cardiac rehabilitation; heart failure; eHealth
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- smartphone-assisted hybrid cardiac rehabilitation (SHCR) (Experimental): Participants receive a 12-wk case manager-led smartphone-assisted hybrid cardiac rehabilitation with follow-up at 12 week and 6 months.
  Interventions: Other: smartphone-assisted hybrid cardiac rehabilitation (SHCR)
- Usual care (No Intervention): Participants receive usual care including general education and exercise suggestion.

INTERVENTIONS:
Other: smartphone-assisted hybrid cardiac rehabilitation (SHCR) — The 12-week case manager-led SHCR program includes:
  * Customized exercise prescriptions following ACSM's heart failure guidelines.
  * A hybrid program combining in-person sessions, home self-exercise, and videoconferencing for exercise coaching(optional), supported by a smartphone app.
  * Case managers instruct patients on a communication app for weekly follow-ups, health education messages, exercise reminders, and progress tracking, including metrics like blood pressure, heart rate, weight, and symptoms.
  Arms: smartphone-assisted hybrid cardiac rehabilitation (SHCR)

SUMMARY:
The aim of this randomized controlled trial is to compare the impact of a case manager-led smartphone-assisted hybrid cardiac rehabilitation program with usual care in patients with HF. Participants will undergo a 12-week program led by a case manager and assisted by a smartphone. The study aims to answer two main questions:

1. Is the novel cardiac rehabilitation model feasible for patients with HF?
2. Does the intervention group show a significant improvement in exercise capacity and adherence compared to the usual care group?

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure between the ages of 18 and 80 years old.
* NYHA (New York Heart Association) functional classification of 1 to 3.
* Patients must be in a stable condition and under outpatient follow-up.

Exclusion Criteria:

* Patients who have contraindications for exercise according to the American College of Sports Medicine's Guidelines for Exercise Testing and Prescription.
* Patients who are unable to complete cardiopulmonary exercise testing.
* Patients who are unable to follow verbal instructions.
* Patients who are unable to walk independently or pedal a stationary bicycle.
* Patients who are unable to use communication app on a smartphone.
* Patients who already engage in physical activity exceeding the recommended moderate intensity of 150 minutes per week or are currently participating in cardiac rehabilitation.
* Patients who do not provide consent to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of peak oxygen uptake | at baseline, 12 weeks(post-intervention), and 6 months.
  Peak oxygen uptake will be assessed using cardiopulmonary exercise test before intervention, at 12 weeks (post-intervention), and at 6 months.
Change of 6 minute walking test | at baseline, 12 weeks(post-intervention), and 6 months.
  6 minute walking test will be performed before intervention, at 12 weeks (post-intervention), and at 6 months.

SECONDARY OUTCOMES:
Adherence to prescribed exercise | 12 weeks(post-intervention)
  We will evaluate the percentage of completed prescribed exercises at 12 weeks.
Evaluation of Quality of life | at baseline, 12 weeks(post-intervention), and 6 months.
  The investigators will assess the change in 36-Item Short Form Survey(SF-36).
Depression | at baseline, 12 weeks(post-intervention), and 6 months.
  The investigators will assess the change in Patient Health Questionnaire (PHQ-9). The PHQ-9 score ranges from 0-27. Higher scores indicate worsen symptoms.
Anxiety | at baseline, 12 weeks(post-intervention), and 6 months.
  The investigators will assess the change in Generalized Anxiety Disorder scale (GAD-7). The GAD-7 score ranges 0-21. Higher scores indicate worsen symptoms.
Evaluation of physical activity | at baseline, 12 weeks(post-intervention), and 6 months.
  The investigators will assess the change in physical activity using International Physical Activity Questionnaire(IPAQ) Taiwan version.
Evaluation of grip strength | at baseline, 12 weeks(post-intervention), and 6 months.
  The grip strength will be measured using a grip goniometer with the participants seated and the elbow flexed at 90 degrees.
Evaluation of frailty | at baseline, 12 weeks(post-intervention), and 6 months.
  The investigators will evaluate the change in the Clinical Frailty Scale, which ranges from 1 to 9. Higher scores represent greater illness.
Blood test: Total cholesterol | at baseline, 12 weeks(post-intervention), and 6 months.
  The Total cholesterol will be tested in the laboratory.
Blood test: LDL | at baseline, 12 weeks(post-intervention), and 6 months.
  The LDL will be tested in the laboratory.
Blood test: HDL | at baseline, 12 weeks(post-intervention), and 6 months.
  The HDL will be tested in the laboratory.
Blood test: Triglyceride | at baseline, 12 weeks(post-intervention), and 6 months.
  The Triglyceride will be tested in the laboratory.
Blood test: NT-proBNP | at baseline, 12 weeks(post-intervention), and 6 months.
  The NT-proBNP will be tested in the laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Jui Chuang, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital, Taipei, Taiwan